CLINICAL TRIAL: NCT05971186
Title: Single-Blinded Randomized Controlled Trial: Comparative Efficacy of Dark Chocolate, Coconut Water, and Ibuprofen in Managing Primary Dysmenorrhea
Brief Title: Dark Chocolate, Coconut Water, and Ibuprofen in Managing Primary Dysmenorrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 703/UN6.KEP/EC/2022
Record Dates: First submitted 2023-07-21; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Dysmenorrhea Primary; Menstrual Pain; Ibuprofen
Keywords: Dark Chocolate; Young Coconut Water; Ibuprofen; Pain Intensity
MeSH Terms: conditions — Dysmenorrhea; Pain | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: The sample comprised 45 female students from Saleha Midwifery Academy who met the inclusion criteria and voluntarily consented after a detailed explanation. Sample size was determined using the Federer formula, yielding a minimum of 9 participants per group. However, 15 samples were included in each of the three treatment groups, resulting in a total of 45 subjects due to the three interventions.
  Simple random sampling via Microsoft Excel's random name selection feature was used to select participants from the accessible population. Random allocation to treatment or control groups was done without bias, using a blocking system and designated application.
  The samples were divided into three groups: Group 1 received young coconut water, Group 2 received 70% dark chocolate bar, and Group 3 received 1 tablet of Ibuprofen, an NSAID. Allocation to each group was randomized using a designated application and a block system.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: This quantitative study uses a Single-blind Randomized Controlled Trial (RCT) design. Key roles, including researcher, subjects, data analyst, collector, and assistant, ensure blinding to individual treatments. Blinding subjects is infeasible due to distinct interventions (young coconut water, dark chocolate, Ibuprofen). The research hypothesis remains undisclosed in the Informed Consent. Subjects won't discuss interventions with involved parties. Implementing this robust design aims to generate unbiased results contributing to scientific knowledge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen (Active Comparator): Fifteen participants were randomly selected to form the third intervention group. Each subject in this arm received a single tablet of Ibuprofen, with a dosage of 400 mg. Similar to the other arms, they were given a 15-minute window to take the Ibuprofen tablet.
  Prior to administering the Ibuprofen, the pain intensity of the participants was measured using the standardized Numeric Rating Scale (NRS). Additionally, the pain intensity was measured again two hours after the consumption of the Ibuprofen tablet, using the same Numeric Rating Scale (NRS).
  Interventions: Drug: Ibuprofen 400 mg
- Young Coconut Water (Active Comparator): Fifteen participants were randomly selected to join the intervention group. Each subject in this arm received a single dose of 330 ml of young coconut water. To ensure uniformity, they were given a 15-minute window to consume the entire 330 ml of the young coconut water intervention.
  Before administering the young coconut water, the pain intensity of the participants was measured using a standardized Numeric Rating Scale (NRS). Additionally, the pain intensity was reevaluated two hours after the consumption of the young coconut water, using the same Numeric Rating Scale (NRS).
  Interventions: Other: Young Coconut Water
- Dark Chocolate Bar (Active Comparator): Fifteen participants were also randomly chosen for the second intervention group. In this arm, each subject received a single 70% dark chocolate bar weighing 35 grams. Similar to Arm 1, they were given a 15-minute timeframe to consume the entire dark chocolate bar intervention.
  Prior to giving the dark chocolate bar, the pain intensity of the participants was measured using the Numeric Rating Scale (NRS). Subsequently, the pain intensity was reassessed two hours after the consumption of the dark chocolate bar, using the same Numeric Rating Scale (NRS).
  Interventions: Other: Dark Chocolate Bar

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Dosage Form: Tablet Dosage: 1 tablet of Ibuprofen (400 mg) Frequency: One-time consumption Duration: Pain intensity measured before consumption and two hours after consumption
  Other Names: Ibuprofen 400 mg - Novapharin
  Arms: Ibuprofen
Other: Young Coconut Water — Dosage Form: Liquid (coconut water) Dosage: 330 ml (milliliters) of young coconut water Frequency: One-time consumption Duration: Pain intensity measured before consumption and two hours after consumption.
  Arms: Young Coconut Water
Other: Dark Chocolate Bar — Dosage Form: Solid (dark chocolate bar) Dosage: 35 grams of 70% dark chocolate Frequency: One-time consumption Duration: Pain intensity measured before consumption and two hours after consumption.
  Arms: Dark Chocolate Bar

SUMMARY:
Dysmenorrhea, the painful condition experienced by women during menstruation, affects a significant proportion of women worldwide and often leads to decreased productivity. Various pharmacological and non-pharmacological treatments are available for pain relief, but information on their effectiveness, particularly regarding green coconut water, dark chocolate, and Ibuprofen, remains limited. This study aimed to compare the effectiveness of green coconut water, dark chocolate bars, and Ibuprofen in reducing the intensity of primary dysmenorrhea. A randomized controlled trial with a quantitative design was conducted, involving 45 participants randomly assigned to receive either 330 ml of green coconut water, 35 grams of 70% dark chocolate, or 400 mg Ibuprofen. Pain intensity was measured before and after treatment.

DETAILED DESCRIPTION:
Dysmenorrhea, commonly known as period pain, is a prevalent condition that affects a large number of women during menstruation, causing discomfort and often leading to reduced productivity. While several treatments are available to alleviate the pain, there is limited information on the comparative effectiveness of different interventions, including green coconut water, dark chocolate, and Ibuprofen.

This research aimed to conduct a randomized controlled trial to compare the effectiveness of green coconut water, dark chocolate bars, and Ibuprofen in managing primary dysmenorrhea. A total of 45 participants were enrolled in the study and randomly assigned to one of three intervention groups: green coconut water, dark chocolate bars, or Ibuprofen.

The green coconut water group received 330 ml of pure green coconut water, which is known for its potential health benefits and natural electrolyte content. The dark chocolate group received 35 grams of 70% dark chocolate, as some studies have suggested its potential role in pain relief due to the presence of bioactive compounds. The Ibuprofen group received 400 mg of the common over-the-counter nonsteroidal anti-inflammatory drug (NSAID) known for its analgesic properties.

To assess the effectiveness of each intervention, pain intensity was measured before and after treatment using validated pain scales. The Kruskal-Wallis test, a non-parametric statistical method, was used to analyze the data and compare the effectiveness of the three interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 17 and 24 years
* Diagnosed with primary dysmenorrhea based on specific characteristics and assessment
* Willing to refrain from using any pharmacological or non-pharmacological therapies other than the interventions provided by the researcher
* willing to participate as respondents

Exclusion Criteria:

* Allergies to dark chocolate or young coconut water or contraindications to Ibuprofen consumption
* Diagnosed with specific gynecological conditions.

Ages: 17 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — In this study, eligibility criteria based on gender require the participation of individuals identifying as female. The research focuses on assessing the effectiveness of interventions for managing primary dysmenorrhea, a condition specific to individuals with female reproductive systems. Therefore, only individuals who identify as female and experience primary dysmenorrhea are eligible to participate in this study. All other gender identities are not included in the eligibility criteria, as the study aims to investigate the impact of the interventions specifically on female participants with primary dysmenorrhea.
Enrollment: 45 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | The Pain intensity measured 2 times. Before the intervention and two hours after the intervention
  Pain intensity was measured using a Numeric Rating Scale (NRS) observation sheet, allowing respondents to rate their pain intensity on a scale from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Kaifar Nuha, STrKeb,M.Keb, Study Director — Universitas Padjadjaran
Locations (1):
- Saleha Academy of Midwifery, Banda Aceh, Special Region of Aceh, Indonesia

REFERENCES:
- [Derived] Nuha K, Rusmil K, Ganiem AR, Permadi W, Diah Herawati DM. Single-Blind Randomized Controlled Trial: Comparative Efficacy of Dark Chocolate, Coconut Water, and Ibuprofen in Managing Primary Dysmenorrhea. Int J Environ Res Public Health. 2023 Aug 21;20(16):6619. doi: 10.3390/ijerph20166619. PMID 37623203